CLINICAL TRIAL: NCT07181707
Title: Correlation Between the Midpalatal Suture Maturity and the Maxillary Third Molar Mineralization: a Cone Beam Computed Tomography Study
Brief Title: Correlation Between the Midpalatal Suture Maturity and the Maxillary Third Molar Mineralization: a CBCT Study
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, VANDE VANNET Bart, Professor, Central Hospital, Nancy, France
Other Study IDs: 2025PI009
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Maturation of the Midpalatal Suture and Maxillary Third Molar Mineralization in Healthy Individuals
Keywords: Molar, third; Cone Beam Computed Tomography; cranial suture; tooth calcification

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patient aged under 14 years: Patients aged under 14 years.
- Patients aged between 14 and 18 years.: Patients aged between 14 and 18 years.
- Patients aged between 19 and 25 years.: Patients aged between 19 and 25 years.
- Patients aged over 25 years.: Patients aged over 25 years.

SUMMARY:
Assessing the maturation of the mid-palatal suture is an essential criterion for orthodontic decision-making. However, from a CBCT according to Angelieri's classification , it remains difficult for the practitioner's untrained eye.

As profile teleradiographs are almost routinely performed in orthodontic check-ups, numerous studies have looked for a correlation between the stage of maturation of the palatal suture and that of the cervical vertebrae. Some have also looked for a link with mineralization of mandibular third or second molars according to Demirjian's classification.

These techniques would provide a reliable and reproducible method without the use of CBCT.

In our study, the investigators will be looking for a correlation with mineralization of the maxillary third molar according to Nolla's classification. The latter has become common in practice and easy to apply on an orthopantomogram.

This would simplify decision-making without the need for a CBCT, but by using the orthopantomogram which is already routinely performed during the assessment.

DETAILED DESCRIPTION:
The study is a non-interventional (observational) research involving the human person, research on existing data (retrospective study).

This study analyzes the maturation stage of the Midpalatal suture and the mineralization of the third left molar.

This is a comparative retrospective study of radiographs in three dimensions before any orthodontic treatment to study a potential correlation.

There is no control group but there are subgroups depending of the age of the patients.

ELIGIBILITY:
Inclusion Criteria:

* No previous orthodontic or orthopedic treatment
* At least the maxillary third left molar
* No skeletal disability

Exclusion Criteria:

* Previous maxillofacial trauma
* Dentofacial deformities
* Endocrinological pathologies with implications for maxillofacial growth • - Syndromes
* History of maxillofacial or orthognathic surgery
* History of orthodontic treatment
* Incomplete data or incomplete CBCT
* Maxillary third left molar fracture/cavity/other deterioratedation

Ages: 9 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Odontology department's patients
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Maturation stages of the midpalatal suture | One day
  Stages according to Angelieri et al.
Third molar calcification | One day
  Calcification's stages of the third left molar maxillary (from 0 to 10) according to Nolla.

CONTACTS AND LOCATIONS:
Overall Officials: Bart VANDE VANNET, PhD, Study Director — Central Hospital, Nancy, France
Locations (1):
- Caroline Bertazzon, Nancy, France, France

IPD SHARING:
Plan to Share IPD: Undecided